CLINICAL TRIAL: NCT06816368
Title: The Thermocool SmartTouch SF Catheter With the Trupulse™ Generator for Endocardial Ablation in Patients With Ventricular Tachycardia
Brief Title: Combined Pulsed Field and Radiofrequency Energy for Ablation of Ventricular Tachycardia
Acronym: DUAL-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Atul Verma, Director of Cardiology, Principal Investigator, Professor of Medicine, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI-CS-020
Record Dates: First submitted 2025-01-25; First posted 2025-02-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Ventricular Tachycardia (V-Tach)
Keywords: ventricular tachycardia; pulsed field ablation; radiofrequency; combined dual energy; catheter ablation; pilot study; human; clinical trial
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation group (Experimental): Patients in this single arm will all undergo clinically-indicated catheter ablation of ventricular tachycardia using a novel combination ablation device capable of delivering both radiofrequency and pulsed field ablation.
  Interventions: Device: Catheter ablation using sequential radiofrequency and pulsed field ablation

INTERVENTIONS:
Device: Catheter ablation using sequential radiofrequency and pulsed field ablation — We are using sequential application of radiofrequency and pulsed field ablation to increase lesion depth and better treat ventricular arrhythmias.

SUMMARY:
This will be a single arm study evaluating a new ablation technology for performing catheter ablation of ventricular tachycardia. The technology combines novel pulsed field ablation with radiofrequency ablation.

DETAILED DESCRIPTION:
One of the limitations of conventional ventricular tachycardia (VT) ablation using radiofrequency (RF) energy is the inability to reach arrhythmogenic tissue deep in the myocardium. Pulsed field (PF) energy, which causes cell death via irreversible electroporation and is non-thermal, may improve outcomes in patients with VT since it has been shown to have better depth penetration in previously scarred tissue. Furthermore, the combination of RF and PF treatment in the same location can increase tissue lesion depth more than either energy alone. This can potentially minimize the need for epicardial ablations, or complex bipolar ablation strategies as well as associated procedural complications. RF and PF have been used extensively for atrial ablation. RF has been the mainstay for all VT ablation but PF use for VT is relatively new.

Pre-clinical work of ventricular ablation procedures in a swine model evaluated the effects of combined and co-localized PF and RF application on cardiac lesion size and their corresponding histological changes. Compared to PF alone ablation, lesion depths and widths were significantly greater in both RF-PF and PF-RF applications. Histology for both combined lesions showed central thermal necrosis surrounded by a hemorrhagic and transitional PF zone. The findings provided evidence for appropriate use of combination therapy in clinical settings.

The design of the study will be carried out as an interventional, prospective, multicenter, single-arm safety and effectiveness evaluation using the Biosense Webster PF/RF Ablation System. The study will enroll subjects with sustained symptomatic VT who are candidates for catheter ablation. Eligible subjects who sign the Informed Consent Form (ICF) and who meet all eligibility criteria will be enrolled and treated with the STSF Catheter in conjunction with the TRUPULSE™ Generator. A maximum sample size of 30 subjects is planned in the study. All study subjects will be followed-up for 6 months after the study procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with two or more documented spontaneous episodes of sustained symptomatic VT within 3 months or 1 sustained episode of VT or VT storm (two or more VTs in 24 hours) which required device therapy (shock or anti-tachycardia pacing), external cardioversion, escalated antiarrhythmic therapy, and / or hospitalization

   * Documented episodes assessment will be performed by a review of ECGs, hospitalization records, and/or Implantable Cardioverter Defibrillator (ICD) interrogation
   * Patients must have an ICD implanted
2. Age ≥18 years
3. LVEF ≥ 30% as estimated by echocardiography, contrast ventriculography, radionuclide imaging or cardiac magnetic resonance imaging within the previous 30 days.
4. Willing and capable of understanding the objective, risk, and requirement of the study, and providing consent.
5. Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria:

1. Definite protruding LV thrombus on pre-ablation imaging.
2. Myocardial infarction (MI) within the preceding 2 months. Patients with incessant VT (present 50% of the time with intervention for a period >12 hrs) may be enrolled if their MI is at least 3 weeks old.
3. Absence of vascular access to the heart chambers.
4. Other disease process likely to limit survival to less than 6 months.
5. Class IV heart failure.
6. Serum creatinine of ≥ 2.5 mg/dl (221 umol/L).
7. Thrombocytopenia (< 50 x 109/L) or coagulopathy.
8. Contraindication to heparin.
9. Women who are pregnant.
10. Cardiac surgery (i.e. ventriculotomy, atriotomy) within the past 2 months. Patients with incessant VT may be enrolled if their surgery is at least 3 weeks old.
11. Acute illness or active systemic infection.
12. Severe aortic stenosis or flail mitral valve.
13. Uncontrolled heart failure.
14. Significant congenital anomaly or medical problem that in the opinion of the principal Investigator would preclude enrollment in the study.
15. Enrolled in an investigational study evaluating another device or drug.
16. Unwilling to participate in the study or unavailable for follow up visits.
17. Previous VT ablation within a year.
18. Epicardial mapping or ablation is anticipated or planned before the VT ablation procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Acute procedural success (elimination of all clinically relevant ventricular tachycardias) | 6 months
  Elimination of all clinically relevant ventricular tachycardias at the end of the procedure.
Primary Safety Outcome | From ablation procedure until 7 days post-ablation
  Primary adverse events (PAE) within 7 days after ablation

SECONDARY OUTCOMES:
Freedom from ventricular tachycardia recurrence at 6 months post-ablation | From ablation until 6 months post-ablation
  Freedom from recurrence (symptomatic or asymptomatic) of monomorphic VT that was targeted at ablation at 6 months following the ablation procedure, plus additional failure modes including acute procedural failure, repeat ablation failure, non-study device failure, AAD failure
Secondary safety outcome | From 7 days until 6 months post-ablation
  Primary adverse events at 7 days - 6 months after ablation

OTHER OUTCOMES:
Quality of life using ICDC score | 6 months post-ablation
  Quality of life using the ICDC quality of life score. There are 20 questions each ranked on a Likert scale from 0 to 4. Points are given for number of questions showing any concern and the degree of concern for a total of 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - IUCPQ, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
All relevant data will be published at study end in final manuscript. This is a small, pilot, first-in-human study.